CLINICAL TRIAL: NCT07082959
Title: The Effect of Nursing Pillow Use on Nipple Pain and Comfort in the Postpartum Period
Brief Title: The Effect of Nursing Pillow Use on Nipple Pain and Comfort
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tuğba Tanrıkulu, Master's Degree Student with Thesis, Istanbul University-Cerrahpasa Midwifery Department, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IUC-SBF-TT-01
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Nipple Pain During Lactation; Comfort
Keywords: Breastfeeding; Nursing pillow; Nipple pain; Comfort; Postpartum period
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Postpartum women will be randomly divided into two groups at a 1:1 ratio, with the intervention group using a breastfeeding pillow, while the control group will not receive any intervention and will continue their routine care.
Masking Description: Due to the visible and practical nature of the intervention (use of a breastfeeding pillow), neither participants nor investigators were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Use of a breastfeeding pillow during the postpartum period to evaluate nipple pain and comfort.
  Interventions: Behavioral: Nursing Pillow
- Control Group (No Intervention): Participants in this group will receive routine postpartum care without a breastfeeding pillow.

INTERVENTIONS:
Behavioral: Nursing Pillow — Although there are studies investigating the effects of breastfeeding pillow use on breastfeeding success, comfort, and positive outcomes for both mother and baby, no study has been found examining the effect of breastfeeding pillow use on nipple pain and maternal comfort in women who have undergone vaginal delivery. Therefore, the aim of this study is to evaluate the effect of breastfeeding pillow use on nipple pain and comfort during the postpartum period.
  Arms: Intervention Group

SUMMARY:
Many factors influence breastfeeding. Nipple pain and comfort are among these factors and can negatively impact the breastfeeding process. A nursing pillow can relieve nipple pain and increase comfort. The purpose of this study was to evaluate the effects of breastfeeding pillow use on nipple pain and comfort.

DETAILED DESCRIPTION:
This study was planned to determine the effect of using a breastfeeding pillow in the postpartum period on nipple pain and maternal comfort. The breastfeeding process is a crucial period not only for ensuring the newborn's adequate nutrition but also for strengthening the bond between mother and baby. The World Health Organization (WHO) and UNICEF recommend initiating breastfeeding within the first hour after birth, exclusively breastfeeding for the first six months, and continuing breastfeeding up to two years of age. However, the sustainability of this process is directly related to the mother's physical comfort and the challenges she encounters.

Nipple pain is one of the most common problems during the breastfeeding period. It is often caused by improper latching of the baby and is one of the leading reasons for early cessation of breastfeeding. Additionally, the mother's inability to maintain a proper body position while breastfeeding may lead to physical discomforts such as back and waist pain, negatively affecting her level of comfort.

In this context, breastfeeding pillows are assistive tools designed to help mothers maintain an appropriate position during breastfeeding, aiming to reduce nipple pain and increase comfort. Although there are studies on the positive effects of breastfeeding pillows on breastfeeding success, comfort, and maternal-infant outcomes, no study has been found that specifically investigates the effect of using a breastfeeding pillow in the postpartum period on nipple pain and maternal comfort in women who had a vaginal delivery.

Therefore, the aim of this study is to evaluate the effect of breastfeeding pillow use during the postpartum period on nipple pain and maternal comfort.

ELIGIBILITY:
Inclusion Criteria:

* Women who gave birth at 37 weeks of gestation or later
* Women who had a vaginal delivery
* Primiparous women
* Women whose babies weigh 2500 grams or more
* Women who are willing to breastfeed their babies
* Women who can speak and understand Turkish

Exclusion Criteria:

* Women who gave birth to twins or more
* Women with previous breastfeeding experience
* Women who experienced postpartum complications
* Women with conditions that may prevent breastfeeding

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2025-08-18 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Nipple Pain | It will be evaluated within the first 24 hours postpartum and on the 7th day.
  The intensity of nipple pain experienced by mothers during breastfeeding measured by Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
Comfort | The Postpartum Comfort Scale is a validated tool consisting of 34 items rated on a 5-point Likert scale. It evaluates physical, psychospiritual, and sociocultural comfort. It will be evaluated within the first 24 hours postpartum and on the 7th day.
  Maternal comfort during breastfeeding assessed using the Postpartum Comfort Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay TÜLAY Yılmaz, Associate Professor, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Cerrahpaşa Faculty of Medicine, Prof. Dr. Murat Dilmener Hospital, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No